CLINICAL TRIAL: NCT02374762
Title: Contact-Free Video Imaging of Arteriovenous Fistulas In Chronic Hemodialysis Patients
Brief Title: Hemodialysis Vascular Access Imaging Study
Status: Completed | Type: Observational
Sponsor: Renal Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15-051
Record Dates: First submitted 2015-02-16; First posted 2015-03-02 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Kidney Disease; Fistula; Hemodialysis Fistula Thrombosis
Keywords: Arteriovenous Fistula; Hemodialysis; Vascular Access
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fistula; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodialysis Patients with AVF: Hemodialysis patients that use an arteriovenous fistula (AVF) to receive their dialysis treatments will be invited to have their AVF recorded by a digital camera for one minute prior to cannulation.

SUMMARY:
The goal of this study is to find the best techniques to take non-invasive images of the arteriovenous fistula (AVF) in hemodialysis patients.

DETAILED DESCRIPTION:
The vascular access is at the same time both the 'lifeline' and the 'Achilles' heel' of hemodialysis patients. Despite improved understanding of the pathophysiology of stenosis and thrombosis of the vascular access, unfortunately translating these advances into either improved therapies or a superior process of care has not been very successful. As a result, there continues to be an epidemic of arteriovenous fistula (AVF) maturation failure, a proliferation of relatively ineffective interventions such as angioplasty and stent placement, an extremely high incidence of catheter use (1).

A major problem is the timely diagnosis of AVF access dysfunction, which - undiagnosed and untreated - will eventually result in its loss. Current methods of diagnosing impending AVF deterioration utilize measurement of access flow, access flow recirculation, ultrasound imaging and angiography. None of these methods are applicable on a per-treatment basis and require some sort of intervention.

Recent advances in video-imaging open the opportunity to non-invasively track AVF movements, possibly on a routine basis. These AVF movements are created by the arterial pulse and routinely checked manually prior to each AVF cannulation. In this research the investigators plan to film the actual AVF movements with the goal to explore the technical feasibility of video-imaging based access surveillance.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years; routinely cannulated AVF in place

Exclusion Criteria:

* inability to communicate in English
* skin maladies which render meaningful AVF imaging impossible
* vascular access procedures in the last 8 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators would like to study patients with chronic kidney disease, currently undergoing hemodialysis via AVF at Renal Research Institute dialysis clinics.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Images of Arteriovenous fistula (AVF) Thrill | 6 months
  To determine if optimized video images can show the movements of the AVF pulse.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kotanko, MD, Principal Investigator — Renal Research Institute
Locations (1):
- Renal Research Institute, New York, New York, United States

REFERENCES:
- [Result] Riella MC, Roy-Chaudhury P. Vascular access in haemodialysis: strengthening the Achilles' heel. Nat Rev Nephrol. 2013 Jun;9(6):348-57. doi: 10.1038/nrneph.2013.76. Epub 2013 Apr 16. PMID 23591442